CLINICAL TRIAL: NCT01648036
Title: Heparin Anticoagulation to Improve Outcomes in Septic Shock: The HALO Pilot
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Ryan Zarychanski, MD MSc. FRCPC, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCA2011/001
Record Dates: First submitted 2012-07-14; First posted 2012-07-24 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Heparin; Dalteparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unfractionated Heparin (Experimental)
  Interventions: Drug: Unfractionated heparin
- Dalteparin (Active Comparator): Standard of care
  Interventions: Drug: Dalteparin

INTERVENTIONS:
Drug: Unfractionated heparin — Dose: 18 IU/kg/hr, continuous intravenous infusion. Duration: up to 7 days or until ICU discharge or death
  Arms: Unfractionated Heparin
Drug: Dalteparin — Dose 5000 IU, subcutaneous, daily
  Other Names: Fragmin
  Arms: Dalteparin

SUMMARY:
Life-threatening infections account for 10% of all intensive care unit admissions and constitute the second more frequent cause of death in the ICU after heart diseases. The most common cause of death in patients admitted with life-threatening infections is multi-organ failure that is mediated by severe inflammation. Given the relationship between inflammation and blood clotting, blood-thinners (also called anticoagulants) have been used to decrease inflammation and the formation of small clots. Several lines of evidence suggest that heparin, a proven and inexpensive blood-thinner, may reduce improve survival in patients diagnosed with life-threatening infection. The primary objective of this study is to demonstrate the feasibility of enrolling patients in a large randomized controlled trial investigating heparin in patients with severe infections. In this study, patients with life-threatening infections will have an equal chance of receiving an intravenous infusion of heparin, or a low dose of a similar drug to prevent of blood clots while patients are immobile. The primary purpose of the study is to demonstrate that an average of 2 patients per site, per month, can be enrolled. Other measures of feasibility include the consent rate, the number of protocol violations that occur during the trial, and the number of dose reductions needed due to excessive anticoagulation. To study the biologic effects of heparin in patients with severe infection, specific laboratory markers will be measured and analyzed. If the feasibility of the trial is confirmed, a large randomized trial designed to tell if heparin can safely improve survival will be conducted. Given its low cost and availability, if heparin is shown to improve survival in patients with severe infection, adoption of this therapy on a global scale is anticipated.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Refractory hypotension documented within 36 hours prior to enrolment that requires institution and ongoing use of vasopressor agents (phenylephrine, norepinephrine, vasopressin, epinephrine, or dopamine > 5 mcg/kg/min) at the time of enrolment. Refractory hypotension is defined as a systolic blood pressure < 90 mmHG or a systolic blood pressure more than 30 mmHg below baseline, or a mean arterial pressure less than 65 mmHG and receipt of greater than or equal to 2 litres of intravenous fluid for the treatment of hypotension.
3. At least 1 other new organ dysfunction defined by the following:

   * Creatinine ≥ 150 µmol/L, or ≥ 1.5x the upper limit of normal or the known baseline creatinine, or < 0.5 ml/kg or urine output for 2 hours(Patients on chronic hemodialysis or peritoneal dialysis must meet one of the following criteria)
   * Need for invasive mechanical ventilation or a P/F ratio < 250
   * Platelets < 100 x109/L, or a drop of 50 x109/L in the 3 days prior to enrollment
   * Arterial pH < 7.30 or base deficit > 5 mmol/L in association with a lactate >/= to 3.0 mmol/L

Exclusion Criteria:

1. Consent declined
2. Clinically apparent other forms of shock including cardiogenic, obstructive (massive pulmonary embolism, cardiac tamponnade, tension pneumothorax), hemorrhagic, neurogenic, or anaphylactic
3. Received vasopressor therapy for greater than 36 hours prior to enrollment
4. Have a significant risk of bleeding as evidenced by one of the following:

   * Clinical: Surgery requiring general or spinal anesthesia within 24 hours prior to enrollment, or the potential need for such surgery in the next 24 hours; evidence of active bleeding; a history of severe head trauma requiring hospitalization; intracranial surgery, or stroke within 3 months before the study or any history of intracerebral arteriovenous malformation, cerebral aneurysm, or mass lesions of the central nervous system; a history of congenital bleeding diatheses; gastrointestinal bleeding within 6 weeks before the study unless corrective surgery had been performed; trauma considered to increase the risk of bleeding; presence of an epidural catheter
   * Laboratory: Platelet count < 30 x109/L, INR > 2.0, or baseline aPTT > 50 sec prior to enrollment.
5. Have an indication for therapeutic anticoagulation (e.g. ACS, acute VTE, mechanical valve, etc)
6. Intent of the most responsible physician to prescribe rhAPC
7. Have had a known or suspected adverse reaction to UFH including HIT
8. Are currently enrolled in related trial
9. Known or suspected cirrhosis, or chronic ascites
10. Use of any of the following medications or treatment regimens: unfractionated heparin to treat an active thrombotic event within 12 hours before the infusion enrollment; low-molecular-weight heparin at a higher dose than recommended for prophylactic use (as specified in the package insert) within 12 hours before the infusion; warfarin (if used within 7 days before study entry AND if the INR time exceeded the upper limit of the normal range for the institution); thrombolytic therapy within 3 days before the study, glycoprotein IIb/IIIa antagonists within 7 days before study entry; protein C or rhAPC within 24 hours before enrollment.
11. Terminal illness with a life expectancy of less than 3 months
12. Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrollment - to enrol an average of 2 patients per site per month over the duration of the study | 1 year
  The primary measure of feasibility is the ability of participating sites to enroll an average of 2 patients per month.

SECONDARY OUTCOMES:
Feasibility(1) - Consent rate - will be considered adequate if 60% of eligible patients are enrolled in the HALO pilot | 1 year
Safety - Rate of major and minor bleeding events | Duration of ICU admission, or up to day +9
  a.) Rates of major and minor bleeding will be adjudicated and will be considered in the context of monitored aPTTs: 1) in the context of aPTTs ≤95 seconds, the rate of major bleeding will be deemed acceptable if major bleeding occurs in ≤10% of patients; and 2) if >20% of patients require an initial (6 hour aPTT) dose reduction of the study drug due to an aPTT >95 seconds, this dose will be deemed infeasible as an initiation dose.
Activation of coagulation - Thrombin-antithrombin (TAT) complexes | Day 1, 2, 3, 5, 7, and 9 (or ICU discharge)
Feasibility(2): Protocol Deviations - The investigators believe that an acceptable rate of protocol violations resulting in a non-scheduled dose reduction or interruption of the study drug to be less than 10% of all study drug dose adjustments | Duration of study drug infusion or up to a maximum of 7 days
Feasibility(3) - Time from randomization to initiation of study drug | the outcome will be assessed during the first 24 hours of enrollment
  The investigators will consider the time from randomization to study treatment initiation to be satisfactory if this interval is less than 4 hours.
Activation of coagulation - Protein C concentration | Day 1, 2, 3, 5, 7, and 9 (or ICU discharge)
Activation of Coagulation - Quantitative d-dimer | Days 1, 2, 3, 5, 7, and 9 (or ICU discharge)
Markers of Inflammation (IL-6, IL-8, IL-10, and IL-17) | Days 1, 2, 3, 5, 7, and 9 (or ICU discharge)
ICU Mortality (Tertiary, descriptive outcome only) | Will be assessed at the time of ICU discharge or death; expected average length of ICU admission is 5.7 days
Hospital Mortality (Tertiary, descriptive outcome only) | Will be assessed at the time of hospital discharge or death; expected average length of hospital admission is 14 days
Change in MODS score (Tertiary, descriptive outcome only) | Will be assessed daily during admission to the ICU; expected average length of ICU admission is 5.7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Zarychanski, MD MSc, Principal Investigator — University of Manitoba; Dean Fergusson, PhD MHA, Principal Investigator — Ottawa Hospital Research Institute
Locations (9):
- Canada (9):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Capital Health - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - St Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Ottawa Hospital Civic Campus, Ottawa, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - Hopital de l'Enfant-Jesus, Québec, Quebec